CLINICAL TRIAL: NCT02505542
Title: A Multicenter, Open-label (Part A) Followed by a Randomized, Double-blind, Parallel-group, Placebo Controlled Study (Part B) to Evaluate Maintenance of Remission in Subjects With Active Axial Spondyloarthritis (axSpA) Receiving Either Certolizumab Pegol 200 mg Q2W or 200 mg Q4W as Compared to Placebo
Brief Title: Study to Evaluate Maintenance of Sustained Remission of axSpA With CZP Compared to Placebo
Acronym: C-OPTIMISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AS0005; 2015-000339-34 (EudraCT Number)
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2015-07-16; First posted 2015-07-22 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Axial Spondyloarthrithis; Ankylosing Spondylitis
Keywords: Axial Spondyloarthritis; axSpA; Ankylosing Spondylitis; Anti TNF-alpha; Certolizumab Pegol; Remission; Spondylarthropathies; Arthritis; Spinal Diseases; Immunosuppressive Agents
MeSH Terms: conditions — Spondylitis, Ankylosing; Axial Spondyloarthritis; Spondylarthropathies; Arthritis; Spinal Diseases | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Open-label Certolizumab Pegol (Other): Certolizumab Pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 6 to Week 48 (Part A). Subjects in sustained remission at Week 48 are eligible for randomization into Part B.
  Interventions: Biological: Certolizumab Pegol
- Double-blind Certolizumab Pegol 200 mg Q2W (Experimental): Certolizumab Pegol (CZP) 200 mg subcutaneous (sc) every 2 weeks (Q2W) from Week 48 onwards.
  Interventions: Biological: Certolizumab Pegol
- Double-blind Certolizumab Pegol 200 mg Q4W (Experimental): Certolizumab Pegol (CZP) 200 mg subcutaneous (sc) every 4 weeks (Q4W) from Week 48 onwards.
  At visits where CZP is not received, subjects receive one injection of Placebo to maintain the study blind.
  Interventions: Biological: Certolizumab Pegol; Other: Placebo
- Placebo (Placebo Comparator): One placebo injection is administered every 2 weeks from Week 48 onwards.
  Interventions: Other: Placebo
- Placebo to CZP 200 mg Q2W escape (Other): Subjects randomized to Placebo who meet flare criteria receive CZP 400 mg subcutaneous (sc) every 2 weeks (Q2W) for the first 3 visits after flare has been confirmed. After that, CZP 200 mg is given every 2 weeks in open-label fashion.
  Interventions: Biological: Certolizumab Pegol; Other: Placebo
- CZP 200 mg Q4W to CZP 200 mg Q2W escape (Other): Subjects randomized to CZP 200 mg Q4W who meet flare criteria receive CZP 200 mg subcutaneous (sc) every 2 weeks (Q2W) for all visits after flare has been confirmed. At the first 3 visits after flare has been confirmed, subjects receive one injection of 200 mg CZP and one injection of Placebo to maintain the study blind.
  Interventions: Biological: Certolizumab Pegol; Other: Placebo
- CZP 200 mg Q2W to CZP 200 mg Q2W escape (Other): Subjects randomized to CZP 200 mg Q2W who meet flare criteria receive CZP 200 mg subcutaneous (sc) every 2 weeks (Q2W) for all visits after flare has been confirmed. At the first 3 visits after flare has been confirmed, subjects receive one injection of 200 mg CZP and one injection of Placebo to maintain the study blind.
  Interventions: Biological: Certolizumab Pegol; Other: Placebo

INTERVENTIONS:
Biological: Certolizumab Pegol — * Active substance: Certolizumab Pegol
  * Pharmaceutical form: Prefilled syringe
  * Concentration: 200 mg / ml
  * Route of Administration: Subcutaneous injection
  Other Names: Cimzia; CDP870
  Arms: CZP 200 mg Q2W to CZP 200 mg Q2W escape; CZP 200 mg Q4W to CZP 200 mg Q2W escape; Double-blind Certolizumab Pegol 200 mg Q2W; Double-blind Certolizumab Pegol 200 mg Q4W; Open-label Certolizumab Pegol; Placebo to CZP 200 mg Q2W escape
Other: Placebo — * Active substance: Placebo
  * Pharmaceutical form: Prefilled syringe
  * Concentration: 0.9 % Saline
  * Route of Administration: Subcutaneous injection
  Arms: CZP 200 mg Q2W to CZP 200 mg Q2W escape; CZP 200 mg Q4W to CZP 200 mg Q2W escape; Double-blind Certolizumab Pegol 200 mg Q4W; Placebo; Placebo to CZP 200 mg Q2W escape

SUMMARY:
Patients receive study drug for one year (Part A). If, after the initial run-in phase, a sustained remission is reached they will be randomly split into one of three dose groups for another year (Part B). The maintenance of the sustained remission will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of adult-onset axial SpondyloArthritis (axSpA) with at least 3 months' symptom duration and meet the Assessment of SpondyloArthritis International Society (ASAS) criteria for axSpA and symptom duration of less than 5 years prior to the participation of this study
* Active disease at Screening as defined by

  * Ankylosing Spondylitis Disease Activity Score (ASDAS) ≥ 2.1
  * Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score ≥ 4
  * Spinal pain > 4 on a 0 to 10 Numerical Rating Scale (NRS) (from BASDAI Item 2)
  * for modified New York (mNY) -negative subjects only: C-reactive Protein (CRP) > upper limit of normal (ULN) and/or current evidence for sacroiliitis on the Screening Magnetic Resonance Imaging (MRI)
* Inadequate response to, or contraindication to, or intolerant to at least 2 Nonsteroidal Anti-Inflammatory Drugs (NSAIDs)

Exclusion Criteria:

* Presence of total Spinal Ankylosis ('bamboo spine')
* Diagnosis of any other Inflammatory Arthritis
* Prior treatment with any experimental biological agents for treatment of Axial SpondyloArthritis (SpA)
* Exposure to more than 1 TNF-antagonist or primary failure to TNF antagonist therapy
* History of or current chronic or recurrent infections
* High risk of infection
* Recent live vaccination
* Concurrent malignancy or a history of malignancy
* Class III or IV congestive heart failure - New York Heart Association (NYHA)
* Demyelinating disease of the central nervous system
* Female subjects who are breastfeeding, pregnant or plan to become pregnant during the study or within 3 months following the last dose of the investigational product
* Subjects with any other condition which, in the investigator's judgment, would make the subject unsuitable for inclusion in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 736 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273(UCB)
Locations (108):
- United States (16):
  - As0005 2313, Glendale, Arizona
  - As0005 2316, Mesa, Arizona
  - As0005 2314, Phoenix, Arizona
  - As0005 2317, Sun City, Arizona
  - As0005 2307, Palm Desert, California
  - As0005 2310, San Francisco, California
  - As0005 2305, Upland, California
  - As0005 2308, Denver, Colorado
  - As0005 2302, Brandon, Florida
  - As0005 2321, Hagerstown, Maryland
  - As0005 2312, Minot, North Dakota
  - As0005 2323, Oklahoma City, Oklahoma
  - As0005 2311, Duncansville, Pennsylvania
  - As0005 2315, Jackson, Tennessee
  - As0005 2303, Austin, Texas
  - As0005 2318, Dallas, Texas
- Belgium (4):
  - As0005 1006, Genk
  - As0005 1001, Ghent
  - As0005 1004, Merksem
  - As0005 1003, Mons
- Bulgaria (7):
  - As0005 1109, Pleven
  - As0005 1103, Plovdiv
  - As0005 1106, Plovdiv
  - As0005 1111, Rousse
  - As0005 1110, Sevlievo
  - As0005 1101, Sofia
  - As0005 1108, Sofia
- Czechia (13):
  - As0005 1308, Brno
  - As0005 1309, Bruntál
  - As0005 1301, Kladno
  - As0005 1307, Ostrava
  - As0005 1303, Pardubice
  - As0005 1302, Prague
  - As0005 1305, Prague
  - As0005 1306, Prague
  - As0005 1310, Prague
  - As0005 1311, Prague
  - As0005 1314, Prague
  - As0005 1313, Uherské Hradiště
  - As0005 1304, Zlín
- France (4):
  - As0005 1504, Montpellier
  - As0005 1505, Orléans
  - As0005 1501, Paris
  - As0005 1503, Tours
- Germany (11):
  - As0005 1406, Berlin
  - As0005 1408, Berlin
  - As0005 1410, Berlin
  - As0005 1412, Berlin
  - As0005 1413, Bochum
  - As0005 1407, Cologne
  - As0005 1405, Erlangen
  - As0005 1404, Frankfurt am Main
  - As0005 1402, Hamburg
  - As0006 1409, Herne
  - As0005 1403, Leipzig
- Hungary (9):
  - As0005 1705, Budapest
  - As0005 1710, Budapest
  - As0005 1704, Debrecen
  - As0005 1706, Miskolc
  - As0005 1711, Nyíregyháza
  - As0005 1707, Szeged
  - As0005 1702, Szentes
  - As0005 1703, Szombathely
  - As0005 1701, Veszprém
- Netherlands (3):
  - As0005 2502, Amsterdam
  - As0005 2503, Rotterdam
  - As0005 2501, Sneek
- Poland (15):
  - As0005 1806, Bialystok
  - As0005 1805, Bydgoszcz
  - As0005 1801, Elblag
  - As0005 1802, Elblag
  - As0005 1812, Krakow
  - As0005 1808, Lodz
  - As0005 1814, Lodz
  - As0005 1803, Lublin
  - As0005 1816, Ostrowiec Świętokrzyski
  - As0005 1809, Poznan
  - As0005 1813, Poznan
  - As0005 1807, Torun
  - As0005 1804, Warsaw
  - As0005 1811, Warsaw
  - As0005 1815, Warsaw
- Romania (8):
  - As0005 1912, Brasov
  - As0005 1904, Brăila
  - As0005 1902, Bucharest
  - As0005 1903, Bucharest
  - As0005 1913, Bucharest
  - As0005 1907, Cluj-Napoca
  - As0005 1910, Iași
  - As0005 1911, Târgu Mureş
- Spain (4):
  - As0005 2403, Córdoba
  - As0005 2404, Getafe
  - As0005 2401, Madrid
  - As0005 2402, Seville
- Taiwan (6):
  - As0005 2205, Kaohsiung City
  - As0005 2201, Taichung
  - As0005 2202, Taichung
  - As0005 2203, Taipei
  - As0005 2204, Taipei
  - As0005 2206, Taipei
- Turkey (Türkiye) (6):
  - As0005 2101, Ankara
  - As0005 2103, Edirne
  - As0005 2102, Gaziantep
  - As0005 2105, Istanbul
  - As0005 2106, Istanbul
  - As0005 2104, Izmir
- United Kingdom (2):
  - As0005 1603, Leeds
  - As0005 1601, Norwich

REFERENCES:
- [Background] Landewe RB, van der Heijde D, Dougados M, Baraliakos X, Van den Bosch FE, Gaffney K, Bauer L, Hoepken B, Davies OR, de Peyrecave N, Thomas K, Gensler LS. Maintenance of clinical remission in early axial spondyloarthritis following certolizumab pegol dose reduction. Ann Rheum Dis. 2020 Jul;79(7):920-928. doi: 10.1136/annrheumdis-2019-216839. Epub 2020 May 7. PMID 32381562
- [Derived] Proft F, Vahldiek JL, Nicolaes J, Tham R, Hoepken B, Ufuktepe B, Poddubnyy D, Bressem KK. Machine learning vs human experts: sacroiliitis analysis from the RAPID-axSpA and C-OPTIMISE phase 3 axSpA trials. Rheumatol Adv Pract. 2025 Apr 18;9(2):rkae118. doi: 10.1093/rap/rkae118. eCollection 2025. PMID 40256636
- [Derived] Baraliakos X, Machado PM, Bauer L, Hoepken B, Kim M, Kumke T, Tham R, Rudwaleit M. Comparison of established and preliminarily proposed ASAS MRI working group cut-offs for inflammatory MRI lesions in the sacroiliac joints in radiographic and non-radiographic axial spondyloarthritis. RMD Open. 2024 Sep 3;10(3):e003886. doi: 10.1136/rmdopen-2023-003886. PMID 39231546
- [Derived] Landewe R, van der Heijde D, Dougados M, Baraliakos X, Van den Bosch F, Gaffney K, Bauer L, Hoepken B, de Peyrecave N, Thomas K, Gensler LS. Induction of Sustained Clinical Remission in Early Axial Spondyloarthritis Following Certolizumab Pegol Treatment: 48-Week Outcomes from C-OPTIMISE. Rheumatol Ther. 2020 Sep;7(3):581-599. doi: 10.1007/s40744-020-00214-7. Epub 2020 Jun 11. PMID 32529495
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in July 2015 and concluded in April 2019.
Pre-assignment Details: The study included 2 parts: Part A with a Screening Period (up to 5 Weeks) and an Open-Label Period (Week 0 to Week 48) and Part B with a Double-Blind Period (Week 48 to Week 96) and a Safety Follow-Up Period (10 weeks after the last dose of study medication).
  Participant Flow refers to the Open-Label Set.
Groups:
- Certolizumab Pegol Open-Label: Participants in this arm received certolizumab pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 6 to Week 48 (Part A). Participants in sustained remission at Week 48 were eligible for randomization into Part B.
- Placebo Double-Blind: Participants in this arm received Placebo subcutaneous (sc) every 2 weeks from Week 48 onwards.
- Certolizumab Pegol 200 mg Q2W Double-Blind: Participants in this arm received certolizumab pegol (CZP) 200 mg subcutaneous (sc) every 2 weeks (Q2W) from Week 48 onwards.
- Certolizumab Pegol 200 mg Q4W Double-Blind: Participants in this arm received certolizumab pegol (CZP) 200 mg subcutaneous (sc) every 4 weeks (Q4W) from Week 48 onwards. At visits where CZP was not received, subjects received one injection of Placebo to maintain the study blind.
Period: Part A: Open-Label Period
Arm/Group | Certolizumab Pegol Open-Label | Placebo Double-Blind | Certolizumab Pegol 200 mg Q2W Double-Blind | Certolizumab Pegol 200 mg Q4W Double-Blind
Started | 736 | 0 | 0 | 0
Completed | 659 | 0 | 0 | 0
Not Completed | 77 | 0 | 0 | 0
Not completed — Adverse Event | 31 | 0 | 0 | 0
Not completed — Lack of Efficacy | 5 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 27 | 0 | 0 | 0
Not completed — New medical history available | 1 | 0 | 0 | 0
Not completed — Participant did not attend week 48 visit | 1 | 0 | 0 | 0
Not completed — Pregnancy | 2 | 0 | 0 | 0
Not completed — Sponsor directive | 1 | 0 | 0 | 0
Not completed — Medical monitor decision | 1 | 0 | 0 | 0
Not completed — Screening failure (detected too late) | 1 | 0 | 0 | 0
Not completed — Non-compliance | 1 | 0 | 0 | 0
Period: Completed Part A, Did Not Enter Part B
Arm/Group | Certolizumab Pegol Open-Label | Placebo Double-Blind | Certolizumab Pegol 200 mg Q2W Double-Blind | Certolizumab Pegol 200 mg Q4W Double-Blind
Started | 659 | 0 | 0 | 0
Completed | 313 | 0 | 0 | 0
Not Completed | 346 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0
Not completed — The subject was not eligible for Part B | 341 | 0 | 0 | 0
Period: Part B: Double-Blind Period
Arm/Group | Certolizumab Pegol Open-Label | Placebo Double-Blind | Certolizumab Pegol 200 mg Q2W Double-Blind | Certolizumab Pegol 200 mg Q4W Double-Blind
Started | 0 | 104 | 104 | 105
Started Escape Period | 0 | 73 | 7 | 15
Completed | 0 | 92 | 95 | 98
Not Completed | 0 | 12 | 9 | 7
Not completed — Adverse Event | 0 | 0 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 8 | 7 | 2
Not completed — Planning pregnancy | 0 | 1 | 0 | 0
Not completed — Week 94 missed | 0 | 0 | 1 | 0
Not completed — Patient was moved from the country | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Miscalculation | 0 | 1 | 0 | 0
Not completed — Subject did not complete all visits | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the The Open-Label Set (OLS) which consisted of all study participants who received at least 1 dose of investigational medicinal product (IMP) in the Open-Label Period of the study (Part A).
Arm/Group | Certolizumab Pegol Open-Label
Number analyzed (Participants) | 736
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 729
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222
  Male | 514
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American indian/alaskan native | 2
  Asian | 38
  Black | 1
  White | 681
  Other/Mixed | 5
  Missing | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Part B Who Did Not Experienced a Flare
Description: A participant was considered to have experienced a flare if the participant had an Ankylosing spondylitis disease activity score (ASDAS) greater or equal to (≥) 2.1 at 2 consecutive visits or an ASDAS greater than (>) 3.5 at any visit during Part B up until Week 96.
  A participant qualified for Part B only if he achieved sustained remission after 48 weeks of Open-Label certolizumab pegol (CZP) treatment. Sustained remission was achieved when a participant had an ASDAS less than (<) 1.3 at Week 32 or Week 36 (if ASDAS < 1.3 at Week 32, it must have been < 2.1 at Week 36; if ASDAS < 2.1 at Week 32, it must have been < 1.3 at Week 36) and an ASDAS < 1.3 at Week 48.
  Missing data were handled using non-response imputation (NRI) methods.
Time Frame: From Week 48 to Week 96
Population: The Randomized Set (RS) consisted of all study participants randomized into Part B of the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo Double-Blind (RS): Participants in this arm received Placebo subcutaneous (sc) every 2 weeks from Week 48 onwards.
  Participants formed the Randomized Set (RS).
- Certolizumab Pegol 200 mg Q2W Double-Blind (RS): Participants in this arm received certolizumab pegol (CZP) 200 mg subcutaneous (sc) every 2 weeks (Q2W) from Week 48 onwards.
  Participants formed the RS.
- Certolizumab Pegol 200 mg Q4W Double-Blind (RS): Participants in this arm received certolizumab pegol (CZP) 200 mg subcutaneous (sc) every 4 weeks (Q4W) from Week 48 onwards. At visits where CZP was not received, subjects received one injection of Placebo to maintain the study blind.
  Participants formed the RS.
Arm/Group | Placebo Double-Blind (RS) | Certolizumab Pegol 200 mg Q2W Double-Blind (RS) | Certolizumab Pegol 200 mg Q4W Double-Blind (RS)
Number analyzed (Participants) | 104 | 104 | 105
percentage of participants | 20.2 [13.0 to 29.2] | 83.7 [75.1 to 90.2] | 79.0 [70.0 to 86.4]
Statistical Analysis 1: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q2W Double-Blind (RS); Odds ratio (and corresponding p-value) resulted from a logistic regression model with factors for treatment, geographic region, and modified New York (mNY) classification for study participants who did not experience a flare. An odds ratio > 1 indicates a study participant on CZP was more likely not to experience a flare than a study participant on placebo. Penalized maximum likelihood approach was used for logistic regression; Test type: Superiority; p < 0.001, Regression, Logistic — A fixed sequence testing procedure was used whereby the second test (CZP 200 mg Q4W vs PBO) was interpreted as statistically significant only if the first test (CZP 200 mg Q2W vs PBO) was significant at the 0.05 level as well; Odds Ratio (OR) = 18.822, 95% CI 2-sided [9.605 to 38.864]
Statistical Analysis 2: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q4W Double-Blind (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 14.069, 95% CI 2-sided [7.395 to 27.955]

2. Secondary Outcome: Percentage of Participants Achieving Sustained Remission at Week 48 in Part A
Description: Sustained remission was achieved when a participant had an ASDAS less than (<) 1.3 at Week 32 or Week 36 (if ASDAS < 1.3 at Week 32, it must have been < 2.1 at Week 36; if ASDAS < 2.1 at Week 32, it must have been < 1.3 at Week 36) and an ASDAS < 1.3 at Week 48.
  Missing data were handled using non-response imputation (NRI) methods.
Time Frame: Week 48
Population: The Open-Label Set (OLS) consisted of all study participants who received at least 1 dose of investigational medicinal product (IMP) in the Open-Label Period of the study (Part A).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Certolizumab Pegol Open-Label (OLS): Participants in this arm received certolizumab pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 6 to Week 48 (Part A). Participants in sustained remission at Week 48 were eligible for randomization into Part B.
  Participants formed the Open-Label Set (OLS).
Arm/Group | Certolizumab Pegol Open-Label (OLS)
Number analyzed (Participants) | 736
percentage of participants | 43.9 [40.3 to 47.6]

3. Secondary Outcome: Percentage of Participants in Ankylosing Spondylitis Disease Activity Score (ASDAS) Disease Activity Categories at Week 48 in Part A
Description: The ASDAS was calculated as the sum of the following components:
  0.121 x Back pain (BASDAI Q2 result) 0.058 x Duration of morning stiffness (BASDAI Q6 result) 0.110 x PGADA (Patient's Global Assessment of Disease Activity) 0.073 x Peripheral pain/swelling (BASDAI Q3 result) 0.579 × (natural logarithm [ln] of the (CRP [mg/L] + 1)) Back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue were all assessed on a numerical scale (0 to 10 units).
  Disease activity was measured by categorical response variables:
  * ASDAS-Inactive Disease (ASDAS-ID): ASDAS < 1.3
  * ASDAS-Moderate Disease (ASDAS-MD): ASDAS ≥ 1.3, < 2.1
  * ASDAS-High Disease activity (ASDAS-HD): ASDAS ≥ 2.1, ≤ 3.5
  * ASDAS-very High Disease activity (ASDAS-vHD): ASDAS > 3.5
  Missing data were handled using last observation carried forward (LOCF) methods.
Time Frame: Week 48
Population: The Open-Label Set (OLS) consisted of all study participants who received at least 1 dose of IMP in the Open-Label Period of the study (Part A).
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol Open-Label (OLS)
Number analyzed (Participants) | 736
percentage of participants
  ASDAS-ID | 52.5
  ASDAS-MD | 22.8
  ASDAS-HD | 18.9
  ASDAS-vHD | 5.9

4. Secondary Outcome: Percentage of Participants in Ankylosing Spondylitis Disease Activity Score (ASDAS) Clinical Improvement Categories at Week 48 in Part A
Description: The ASDAS was calculated as the sum of the following components:
  0.121 x Back pain (BASDAI Q2 result) 0.058 x Duration of morning stiffness (BASDAI Q6 result) 0.110 x PGADA (Patient's Global Assessment of Disease Activity) 0.073 x Peripheral pain/swelling (BASDAI Q3 result) 0.579 × (natural logarithm [ln] of the (CRP [mg/L] + 1)) Back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue were all assessed on a numerical scale (0 to 10 units).
  ASDAS improvement was measured by binary response variables:
  * ASDAS-CII: ASDAS reduction (improvement) of ≥ 1.1 relative to Baseline
  * ASDAS-MI: ASDAS reduction (improvement) of ≥ 2.0 relative to Baseline
  Missing data were handled using non-response imputation (NRI) methods.
Time Frame: Week 48
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol Open-Label (OLS)
Number analyzed (Participants) | 736
percentage of participants
  ASDAS-CII | 76.6
  ASDAS-MI | 56.1

5. Secondary Outcome: Time to Flare in Part B
Description: For those who met the criteria for flare (see primary efficacy variable), the time to flare was the length in days from randomization in Part B until the visit at which the criteria for flare were met. Participants who discontinued the study without meeting the criteria for flare were counted as experiencing a flare at the time of their last study visit.
  The time to flare was analyzed using Kaplan-Meier methods. If Kaplan-Meier Estimate was NA for all estimates then more than 75 % failed to meet the flare condition.
  Missing data were handled using non-response imputation (NRI) methods.
Time Frame: From Week 48 to Week 96
Population: The Randomized Set (RS) consisted of all study participants randomized into Part B of the study.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo Double-Blind (RS) | Certolizumab Pegol 200 mg Q2W Double-Blind (RS) | Certolizumab Pegol 200 mg Q4W Double-Blind (RS)
Number analyzed (Participants) | 104 | 104 | 105
days | 113 [84 to 257] | 371 [371 to 371] | NA [NA to NA] — Values were not calculated since more than 75 % failed to meet the flare condition.
Statistical Analysis 1: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q2W Double-Blind (RS); P-values were from stratified log-rank test comparing the Certolizumab pegol 200 mg Q2W Double-Blind (RS) group with the Placebo Double-Blind (RS) group (Geographic region and modified New York (mNY) classification were used as stratification factors); Test type: Other; p < 0.001, Log Rank
Statistical Analysis 2: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q4W Double-Blind (RS); P-values were from stratified log-rank test comparing the Certolizumab pegol 200 mg Q4W Double-Blind (RS) group with the Placebo Double-Blind (RS) group (Geographic region and modified New York (mNY) classification were used as stratification factors); Test type: Other; p < 0.001, Log Rank

6. Secondary Outcome: Percentage of Participants in Ankylosing Spondylitis Disease Activity Score (ASDAS) Disease Activity Categories at Week 96 in Part B
Description: The ASDAS was calculated as the sum of the following components:
  0.121 x Back pain (BASDAI Q2 result) 0.058 x Duration of morning stiffness (BASDAI Q6 result) 0.110 x PGADA (Patient's Global Assessment of Disease Activity) 0.073 x Peripheral pain/swelling (BASDAI Q3 result) 0.579 × (natural logarithm [ln] of the (CRP [mg/L] + 1)) Back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue were all assessed on a numerical scale (0 to 10 units).
  Disease activity was measured by categorical response variables:
  * ASDAS-Inactive Disease (ASDAS-ID): ASDAS < 1.3
  * ASDAS-Moderate Disease (ASDAS-MD): ASDAS ≥ 1.3, < 2.1
  * ASDAS-High Disease activity (ASDAS-HD): ASDAS ≥ 2.1, ≤ 3.5
  * ASDAS-very High Disease activity (ASDAS-vHD): ASDAS > 3.5
Time Frame: Week 96
Population: The Randomized Set (RS) consisted of all study participants randomized into Part B of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Double-Blind (RS) | Certolizumab Pegol 200 mg Q2W Double-Blind (RS) | Certolizumab Pegol 200 mg Q4W Double-Blind (RS)
Number analyzed (Participants) | 104 | 104 | 105
percentage of participants
  ASDAS-ID | 58.3 | 86.2 | 69.9
  ASDAS-MD | 25.0 | 13.8 | 22.9
  ASDAS-HD | 16.7 | 0 | 7.2
  ASDAS-vHD | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants in Ankylosing Spondylitis Disease Activity Score (ASDAS) Clinical Improvement Categories at Week 96 in Part B
Description: as for outcome 4
Time Frame: Week 96
Population: The Randomized Set (RS) consisted of all study participants randomized into Part B of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Double-Blind (RS) | Certolizumab Pegol 200 mg Q2W Double-Blind (RS) | Certolizumab Pegol 200 mg Q4W Double-Blind (RS)
Number analyzed (Participants) | 104 | 104 | 105
percentage of participants
  ASDAS-CII | 21.2 | 82.7 | 75.2
  ASDAS-MI | 10.6 | 67.3 | 58.1
Statistical Analysis 1: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q2W Double-Blind (RS); Odds ratios (and corresponding p-values) were from a logistic regression model with factors for treatment group, geographical region, and modified New York (mNY) classification; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 17.940, 95% CI 2-sided [8.950 to 35.961]
Statistical Analysis 2: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q4W Double-Blind (RS); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 11.385, 95% CI 2-sided [5.952 to 21.778]
Statistical Analysis 3: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q2W Double-Blind (RS); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 17.653, 95% CI 2-sided [8.333 to 37.399]
Statistical Analysis 4: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q4W Double-Blind (RS); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 11.863, 95% CI 2-sided [5.670 to 24.822]

8. Secondary Outcome: Percentage of Participants With Axial SpondyloArthritis International Society 20 % Response Criteria (ASAS20) Response at Week 96 in Part B
Description: The ASAS20 response was defined as an improvement of at least 20 % and absolute improvement of at least 1 unit on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and absence of deterioration in the potential remaining domain [deterioration was defined as a relative worsening of at least 20 % and an absolute worsening of at least 1 unit].
  Missing data were handled using non-response imputation (NRI) methods.
Time Frame: Week 96
Population: The Randomized Set (RS) consisted of all study participants randomized into Part B of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Double-Blind (RS) | Certolizumab Pegol 200 mg Q2W Double-Blind (RS) | Certolizumab Pegol 200 mg Q4W Double-Blind (RS)
Number analyzed (Participants) | 104 | 104 | 105
percentage of participants | 23.1 | 85.6 | 78.1
Statistical Analysis 1: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q2W Double-Blind (RS); Odds ratios (and corresponding p-values) were from a logistic regression model with factors for treatment group, geographical region, and mNY classification; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 20.205, 95% CI 2-sided [9.851 to 41.439]
Statistical Analysis 2: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q4W Double-Blind (RS); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 12.070, 95% CI 2-sided [6.275 to 23.218]

9. Secondary Outcome: Percentage of Participants With Axial SpondyloArthritis International Society 40 % Response Criteria (ASAS40) Response at Week 96 in Part B
Description: The ASAS40 response was defined as a relative improvement of at least 40 % and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and no worsening at all in the remaining domain.
  Missing data were handled using non-response imputation (NRI) methods.
Time Frame: Week 96
Population: The Randomized Set (RS) consisted of all study participants randomized into Part B of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Double-Blind (RS) | Certolizumab Pegol 200 mg Q2W Double-Blind (RS) | Certolizumab Pegol 200 mg Q4W Double-Blind (RS)
Number analyzed (Participants) | 104 | 104 | 105
percentage of participants | 21.2 | 84.6 | 73.3
Statistical Analysis 1: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q2W Double-Blind (RS); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 20.891, 95% CI 2-sided [10.210 to 42.744]
Statistical Analysis 2: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q4W Double-Blind (RS); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 10.377, 95% CI 2-sided [5.456 to 19.738]

10. Secondary Outcome: Percentage of Participants With Axial SpondyloArthritis International Society (ASAS) 5/6 Response Criteria Response at Week 96 in Part B
Description: The ASAS 5/6 response was defined as achieving at least 20 % improvement in 5 of 6 domains, including the 4 domains defined for ASAS20 as well as spinal mobility (lateral spinal flexion) and C-reactive Protein (CRP).
  Missing data were handled using non-response imputation (NRI) methods.
Time Frame: Week 96
Population: The Randomized Set (RS) consisted of all study participants randomized into Part B of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Double-Blind (RS) | Certolizumab Pegol 200 mg Q2W Double-Blind (RS) | Certolizumab Pegol 200 mg Q4W Double-Blind (RS)
Number analyzed (Participants) | 104 | 104 | 105
percentage of participants | 12.5 | 70.2 | 62.9
Statistical Analysis 1: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q2W Double-Blind (RS); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 16.900, 95% CI 2-sided [8.211 to 34.785]
Statistical Analysis 2: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q4W Double-Blind (RS); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 12.072, 95% CI 2-sided [5.954 to 24.476]

11. Secondary Outcome: Percentage of Participants With Axial SpondyloArthritis International Society (ASAS) Partial Remission (PR) Response Criteria Response at Week 96 in Part B
Description: The ASAS partial remission (PR) response was defined as a score of ≤ 2 units on a 0 to 10 unit scale in all 4 domains listed for ASAS20.
  Missing data were handled using non-response imputation (NRI) methods.
Time Frame: Week 96
Population: The Randomized Set (RS) consisted of all study participants randomized into Part B of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Double-Blind (RS) | Certolizumab Pegol 200 mg Q2W Double-Blind (RS) | Certolizumab Pegol 200 mg Q4W Double-Blind (RS)
Number analyzed (Participants) | 104 | 104 | 105
percentage of participants | 17.3 | 77.9 | 70.5
Statistical Analysis 1: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q2W Double-Blind (RS); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 17.082, 95% CI 2-sided [8.561 to 34.085]
Statistical Analysis 2: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q4W Double-Blind (RS); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 11.503, 95% CI 2-sided [5.939 to 22.278]

12. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at Week 96 in Part B
Description: The ASDAS was calculated as the sum of the following components:
  0.121 x Back pain (BASDAI Q2 result) 0.058 x Duration of morning stiffness (BASDAI Q6 result) 0.110 x PGADA (Patient's Global Assessment of Disease Activity) 0.073 x Peripheral pain/swelling (BASDAI Q3 result) 0.579 × (natural logarithm [ln] of the (CRP [mg/L] + 1)) Back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue were all assessed on a numerical scale (0 to 10 units).
  There is a minimum score of 0.636 for the total ASDAS score, but no defined upper score. Based on the formula even in the situation that the CRP is normal, any value below 4 is recorded as "below the limit of quantification" (BLQ) and a value of BLQ/2=2 was prespecified. This assumption is triggering the lowest possible value of 0.636.
  The change from Part B Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Week 48 to Week 96
Population: The Randomized Set (RS) consisted of all study participants randomized into Part B of the study.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo Double-Blind (RS) | Certolizumab Pegol 200 mg Q2W Double-Blind (RS) | Certolizumab Pegol 200 mg Q4W Double-Blind (RS)
Number analyzed (Participants) | 104 | 104 | 105
scores on a scale | 1.66 (0.110) | 0.24 (0.077) | 0.45 (0.077)
Statistical Analysis 1: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q2W Double-Blind (RS); An mixed model with repeated measures (MMRM) analysis on all observed post-baseline data with the following fixed-effect covariates was used: treatment, geographical region, mNY classification, Part B Baseline value, and visit as fixed-effect factors, as well as treatment group by visit interaction and Part B Baseline value by visit interaction; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference vs Placebo = -1.42, 95% CI 2-sided [-1.66 to -1.17], Standard Error of Mean 0.126
Statistical Analysis 2: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q4W Double-Blind (RS); [analysis description as in outcome 12, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference vs Placebo = -1.21, 95% CI 2-sided [-1.45 to -0.96], Standard Error of Mean 0.126

13. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 96 in Part B
Description: The BASDAI is a validated self-reported instrument, which consists of six 10 unit horizontal Numeric Rating Scales (NRS) to measure the disease activity of ankylosing spondylitis (AS) from the subject's perspective. It measures the severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration) over the last week. The final BASDAI scores ranges from 0 to 10, with lower scores indicating lower disease activity.
  The change from Part B Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Week 48 to Week 96
Population: The Randomized Set (RS) consisted of all study participants randomized into Part B of the study.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo Double-Blind (RS) | Certolizumab Pegol 200 mg Q2W Double-Blind (RS) | Certolizumab Pegol 200 mg Q4W Double-Blind (RS)
Number analyzed (Participants) | 104 | 104 | 105
scores on a scale | 3.02 (0.226) | 0.56 (0.176) | 0.78 (0.176)
Statistical Analysis 1: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q2W Double-Blind (RS); [analysis description as in outcome 12, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference vs Placebo = -2.46, 95% CI 2-sided [-2.99 to -1.94], Standard Error of Mean 0.268
Statistical Analysis 2: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q4W Double-Blind (RS); [analysis description as in outcome 12, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference vs Placebo = -2.24, 95% CI 2-sided [-2.77 to -1.72], Standard Error of Mean 0.267

14. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 96 in Part B
Description: The BASFI is a validated disease-specific instrument for assessing physical function. The BASFI comprises 10 items relating to the past week. The BASFI is the mean of the 10 scores such that the total score ranges from 0 (Easy) to 10 (Impossible), with lower scores indicating better physical function.
  The change from Part B Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Week 48 to Week 96
Population: The Randomized Set (RS) consisted of all study participants randomized into Part B of the study.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo Double-Blind (RS) | Certolizumab Pegol 200 mg Q2W Double-Blind (RS) | Certolizumab Pegol 200 mg Q4W Double-Blind (RS)
Number analyzed (Participants) | 104 | 104 | 105
scores on a scale | 1.90 (0.233) | 0.32 (0.198) | 0.46 (0.205)
Statistical Analysis 1: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q2W Double-Blind (RS); [analysis description as in outcome 12, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference vs Placebo = -1.57, 95% CI 2-sided [-2.04 to -1.11], Standard Error of Mean 0.238
Statistical Analysis 2: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q4W Double-Blind (RS); [analysis description as in outcome 12, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference vs Placebo = -1.43, 95% CI 2-sided [-1.90 to -0.96], Standard Error of Mean 0.238

15. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) at Week 96 in Part B
Description: The BASMI is a disease-specific measure consisting of 5 clinical measures to reflect subject axial status: cervical rotation; tragus to wall distance; lateral lumbar flexion; lumbar flexion (modified Schober test); intermalleolar distance. According to the linear definition of the BASMI a score of 0 to 10 was calculated for each item based on the measurement. The mean of the sum of the 5 scores provided the total BASMI score, ranging from 0 to 10. The higher the BASMI score the more severe the patient's limitation of movement due to their axial spondyloarthritis (axSpA).
  The change from Part B Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Week 48 to Week 96
Population: The Randomized Set (RS) consisted of all study participants randomized into Part B of the study.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo Double-Blind (RS) | Certolizumab Pegol 200 mg Q2W Double-Blind (RS) | Certolizumab Pegol 200 mg Q4W Double-Blind (RS)
Number analyzed (Participants) | 104 | 104 | 105
scores on a scale | 0.21 (0.105) | 0.00 (0.065) | -0.03 (0.068)
Statistical Analysis 1: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q2W Double-Blind (RS); [analysis description as in outcome 12, analysis 1]; Test type: Other; p = 0.074, Mixed Models Analysis; LS Mean Difference vs Placebo = -0.20, 95% CI 2-sided [-0.42 to 0.02], Standard Error of Mean 0.112
Statistical Analysis 2: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q4W Double-Blind (RS); [analysis description as in outcome 12, analysis 1]; Test type: Other; p = 0.036, Mixed Models Analysis; LS Mean Difference vs Placebo = -0.24, 95% CI 2-sided [-0.46 to -0.02], Standard Error of Mean 0.113

16. Secondary Outcome: Percentage of Participants With Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 Response Criteria Response at Week 96 in Part B
Description: The BASDAI50 response was defined as an improvement of at least 50 % in the BASDAI score relative to Baseline.
  Missing data were handled using non-response imputation (NRI) methods.
Time Frame: Week 96
Population: The Randomized Set (RS) consisted of all study participants randomized into Part B of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Double-Blind (RS) | Certolizumab Pegol 200 mg Q2W Double-Blind (RS) | Certolizumab Pegol 200 mg Q4W Double-Blind (RS)
Number analyzed (Participants) | 104 | 104 | 105
percentage of participants | 22.1 | 83.7 | 77.1
Statistical Analysis 1: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q2W Double-Blind (RS); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 18.308, 95% CI 2-sided [9.084 to 36.898]
Statistical Analysis 2: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q4W Double-Blind (RS); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 12.020, 95% CI 2-sided [6.255 to 23.098]

17. Secondary Outcome: Change From Baseline in Sacroiliac Spondyloarthritis Research Consortium of Canada (SPARCC) Score at Week 96 in Part B
Description: The SPARCC scoring method for lesions found on the Magnetic Resonance Imaging (MRI) is based on an abnormal increased signal on the Short-Tau-Inversion Recovery (STIR) sequence, representing bone marrow edema. Total Sacroiliac (SI) joint SPARCC score can range from 0 to 72 with higher scores indicating higher joint inflammation.
  The change from Part B Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Week 48 to Week 96
Population: The Randomized Set (RS) consisted of all study participants randomized into Part B of the study.
  The number of participants analyzed reflects Week 96.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo Double-Blind (RS) | Certolizumab Pegol 200 mg Q2W Double-Blind (RS) | Certolizumab Pegol 200 mg Q4W Double-Blind (RS)
Number analyzed (Participants) | 24 | 79 | 77
scores on a scale | 1.1 (3.6) | 0.2 (2.4) | 0.6 (3.8)
Statistical Analysis 1: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q2W Double-Blind (RS); Only MRIs performed ± 2 weeks around the Week 96 or Early Withdrawal Visit were assigned to Week 96 or Early Withdrawal. Only results of the double-read assessments of the central MRI review were included. The analysis used the average of the scores from the 2 independent reviewers. Whenever an adjudication was present, the average score across all 3 reviewers was used. ANCOVA model with treatment, geographical region, mNY classification, and Part B Baseline as covariates; Test type: Other; p = 0.195, ANCOVA; LS Mean Difference vs Placebo = -1.0, 95% CI 2-sided [-2.50 to 0.51], Standard Error of Mean 0.76
Statistical Analysis 2: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q4W Double-Blind (RS); [analysis description as in outcome 17, analysis 1]; Test type: Other; p = 0.432, ANCOVA; LS Mean Difference vs Placebo = -0.6, 95% CI 2-sided [-2.11 to 0.91], Standard Error of Mean 0.76

18. Secondary Outcome: Change From Baseline in Spine Ankylosing Spondylitis Spine Magnetic Resonance Imaging Score for Disease Activity (ASspIMRI-a) in the Berlin Modification Score at Week 96 in Part B
Description: The Berlin modification of the ASspiMRI-a is a scoring system with a concentration on Short-Tau-Inversion Recovery (STIR) sequences without other fat saturation techniques. It quantifies changes in 23 Vertebral Units (VU) of the spine. Active inflammation was scored by grading the degree of bone marrow edema from 0 to 3 in 1 dimension on 1 or more consecutive slices that represent the highest level of inflammation in a particular VU.
  The change from Part B Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Week 48 to Week 96
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo Double-Blind (RS) | Certolizumab Pegol 200 mg Q2W Double-Blind (RS) | Certolizumab Pegol 200 mg Q4W Double-Blind (RS)
Number analyzed (Participants) | 24 | 79 | 78
scores on a scale | 0.4 (0.9) | 0.0 (0.8) | 0.0 (0.8)
Statistical Analysis 1: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q2W Double-Blind (RS); [analysis description as in outcome 17, analysis 1]; Test type: Other; p = 0.040, ANCOVA; LS Mean Difference vs Placebo = -0.4, 95% CI 2-sided [-0.78 to -0.02], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: Placebo Double-Blind (RS) vs Certolizumab Pegol 200 mg Q4W Double-Blind (RS); [analysis description as in outcome 17, analysis 1]; Test type: Other; p = 0.074, ANCOVA; LS Mean Difference vs Placebo = -0.3, 95% CI 2-sided [-0.73 to 0.03], Standard Error of Mean 0.19

19. Secondary Outcome: Percentage of Participants in Ankylosing Spondylitis Disease Activity Score (ASDAS) Disease Activity Categories at Escape Week 12 for Participants Who Experienced a Flare in Part B
Description: as for outcome 6
Time Frame: Escape Week 12
Population: The Flared Set (FS) consisted of all study participants from the RS who experienced a flare in Part B.
Measure: Number; unit: percentage of participants
Groups:
- Placebo DB/CZP 200 mg Q2W Escape (FS): Participants randomized to Placebo who met flare criteria received CZP 400 mg subcutaneous (sc) every 2 weeks (Q2W) for the first 3 visits after flare has been confirmed. After that, CZP 200 mg was given every 2 weeks in open-label fashion. The duration was from starting escape treatment after flare until Week 96 with a minimum of 12 weeks.
  Participants formed the Flared Set (FS).
- CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (FS): Participants randomized to CZP 200 mg Q2W who meet flare criteria received CZP 200 mg subcutaneous (sc) every 2 weeks (Q2W) for all visits after flare has been confirmed. At the first 3 visits after flare has been confirmed, participants received one injection of 200 mg CZP and one injection of Placebo to maintain the study blind. The duration was from starting escape treatment after flare until Week 96 with a minimum of 12 weeks.
  Participants formed the FS.
- CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (FS): Participants randomized to CZP 200 mg Q4W who meet flare criteria received CZP 200 mg subcutaneous (sc) every 2 weeks (Q2W) for all visits after flare has been confirmed. At the first 3 visits after flare has been confirmed, participants received one injection of 200 mg CZP and one injection of Placebo to maintain the study blind. The duration was from starting escape treatment after flare until Week 96 with a minimum of 12 weeks.
  Participants formed the FS.
Arm/Group | Placebo DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (FS)
Number analyzed (Participants) | 73 | 7 | 15
percentage of participants
  ASDAS-ID | 63.4 | 16.7 | 60.0
  ASDAS-MD | 26.8 | 50.0 | 20.0
  ASDAS-HD | 8.5 | 33.3 | 20.0
  ASDAS-vHD | 1.4 | 0 | 0

20. Secondary Outcome: Percentage of Participants in Ankylosing Spondylitis Disease Activity Score (ASDAS) Clinical Improvement Categories at Escape Week 12 for Participants Who Experienced a Flare in Part B
Description: The ASDAS was calculated as the sum of the following components:
  0.121 x Back pain (BASDAI Q2 result) 0.058 x Duration of morning stiffness (BASDAI Q6 result) 0.110 x PGADA (Patient's Global Assessment of Disease Activity) 0.073 x Peripheral pain/swelling (BASDAI Q3 result) 0.579 × (natural logarithm [ln] of the (CRP [mg/L] + 1)) Back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue were all assessed on a numerical scale (0 to 10 units).
  ASDAS improvement was measured by binary response variables:
  * ASDAS-CII: ASDAS reduction (improvement) of ≥ 1.1 relative to Baseline
  * ASDAS-MI: ASDAS reduction (improvement) of ≥ 2.0 relative to Baseline
Time Frame: Escape Week 12
Population: The Flared Set (FS) consisted of all study participants from the RS who experienced a flare in Part B.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (FS)
Number analyzed (Participants) | 73 | 7 | 15
percentage of participants
  ASDAS-CII | 84.5 | 16.7 | 46.7
  ASDAS-MI | 49.3 | 0 | 13.3

21. Secondary Outcome: Percentage of Participants With Axial SpondyloArthritis International Society 20 % Response Criteria (ASAS20) Response at Escape Week 12 for Participants Who Experienced a Flare in Part B
Description: The ASAS20 response was defined as an improvement of at least 20 % and absolute improvement of at least 1 unit on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and absence of deterioration in the potential remaining domain [deterioration was defined as a relative worsening of at least 20% and an absolute worsening of at least 1 unit].
Time Frame: Escape Week 12
Population: The Flared Set (FS) consisted of all study participants from the RS who experienced a flare in Part B.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (FS)
Number analyzed (Participants) | 73 | 7 | 15
percentage of participants | 83.3 | 50.0 | 64.3

22. Secondary Outcome: Percentage of Participants With Axial SpondyloArthritis International Society 40 % Response Criteria (ASAS40) Response at Escape Week 12 for Participants Who Experienced a Flare in Part B
Description: The ASAS40 response was defined as a relative improvement of at least 40 % and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and no worsening at all in the remaining domain.
Time Frame: Escape Week 12
Population: The Flared Set (FS) consisted of all study participants from the RS who experienced a flare in Part B.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (FS)
Number analyzed (Participants) | 73 | 7 | 15
percentage of participants | 69.4 | 16.7 | 50.0

23. Secondary Outcome: Percentage of Participants With Axial SpondyloArthritis International Society (ASAS) 5/6 Response Criteria Response at Escape Week 12 for Participants Who Experienced a Flare in Part B
Description: The ASAS 5/6 response was defined as achieving at least 20 % improvement in 5 of 6 domains, including the 4 domains defined for ASAS20 as well as spinal mobility (lateral spinal flexion) and C-reactive Protein (CRP).
Time Frame: Escape Week 12
Population: The Flared Set (FS) consisted of all study participants from the RS who experienced a flare in Part B.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (FS)
Number analyzed (Participants) | 73 | 7 | 15
percentage of participants | 60.6 | 16.7 | 7.1

24. Secondary Outcome: Percentage of Participants With Axial SpondyloArthritis International Society (ASAS) Partial Remission (PR) Response Criteria Response at Escape Week 12 for Participants Who Experienced a Flare in Part B
Description: The ASAS partial remission (PR) response was defined as a score of ≤ 2 units on a 0 to 10 unit scale in all 4 domains listed for ASAS20.
Time Frame: Escape Week 12
Population: The Flared Set (FS) consisted of all study participants from the RS who experienced a flare in Part B.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (FS)
Number analyzed (Participants) | 73 | 7 | 15
percentage of participants | 66.7 | 16.7 | 50.0

25. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at Escape Week 12 for Participants Who Experienced a Flare in Part B
Description: as for outcome 12
Time Frame: From time of flare to Escape Week 12
Population: The Flared Set (FS) consisted of all study participants from the RS who experienced a flare in Part B.
  The number of participants analyzed reflects Escape Week 12.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (FS)
Number analyzed (Participants) | 71 | 6 | 15
scores on a scale | -2.18 (1.13) | -0.56 (0.64) | -0.83 (0.94)

26. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Escape Week 12 for Participants Who Experienced a Flare in Part B
Description: The BASDAI is a validated self-reported instrument, which consists of six 10 unit horizontal Numeric Rating Scales (NRS) to measure the disease activity of ankylosing spondylitis (AS) from the subject's perspective. It measures the severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration) over the last week. The final BASDAI scores ranges from 0 to 10, with lower scores indicating lower disease activity.
  The change from flare Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From time of flare to Escape Week 12
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (FS)
Number analyzed (Participants) | 72 | 6 | 15
scores on a scale | -3.75 (2.52) | -1.55 (1.05) | -2.29 (2.35)

27. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Escape Week 12 for Participants Who Experienced a Flare in Part B
Description: The BASFI is a validated disease-specific instrument for assessing physical function. The BASFI comprises 10 items relating to the past week. The BASFI is the mean of the 10 scores such that the total score ranges from 0 (Easy) to 10 (Impossible), with lower scores indicating better physical function.
  The change from flare Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From time of flare to Escape Week 12
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (FS)
Number analyzed (Participants) | 72 | 6 | 14
scores on a scale | -2.52 (2.46) | -0.72 (0.70) | -1.83 (2.38)

28. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) at Escape Week 12 for Participants Who Experienced a Flare in Part B
Description: The BASMI is a disease-specific measure consisting of 5 clinical measures to reflect subject axial status: cervical rotation; tragus to wall distance; lateral lumbar flexion; lumbar flexion (modified Schober test); intermalleolar distance. According to the linear definition of the BASMI a score of 0 to 10 was calculated for each item based on the measurement. The mean of the sum of the 5 scores provided the total BASMI score, ranging from 0 to 10. The higher the BASMI score the more severe the patient's limitation of movement due to their axial spondyloarthritis (axSpA).
  The change from flare Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From time of flare to Escape Week 12
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (FS)
Number analyzed (Participants) | 67 | 6 | 15
scores on a scale | -0.43 (0.58) | -0.27 (0.35) | -0.26 (0.30)

29. Secondary Outcome: Change From Baseline in Sacroiliac Spondyloarthritis Research Consortium of Canada (SPARCC) Score at Escape Week 12 for Participants Who Experienced a Flare in Part B
Description: The SPARCC scoring method for lesions found on the Magnetic Resonance Imaging (MRI) is based on an abnormal increased signal on the Short-Tau-Inversion Recovery (STIR) sequence, representing bone marrow edema. Total Sacroiliac (SI) joint SPARCC score can range from 0 to 72 with higher scores indicating higher joint inflammation.
  The change from flare Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From time of flare to Escape Week 12
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (FS)
Number analyzed (Participants) | 48 | 2 | 12
scores on a scale | -9.3 (13.2) | 0.0 (0.0) | 0.2 (3.1)

30. Secondary Outcome: Change From Baseline in Spine Ankylosing Spondylitis Spine Magnetic Resonance Imaging Score for Activity (ASspIMRI-a) in the Berlin Modification Score at Escape Week 12 for Participants Who Experienced a Flare in Part B
Description: The Berlin modification of the ASspiMRI-a is a scoring system with a concentration on Short-Tau-Inversion Recovery (STIR) sequences without other fat saturation techniques. It quantifies changes in 23 Vertebral Units (VU) of the spine. Active inflammation was scored by grading the degree of bone marrow edema from 0 to 3 in 1 dimension on 1 or more consecutive slices that represent the highest level of inflammation in a particular VU.
  The change from flare Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From time of flare to Escape Week 12
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (FS) | CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (FS)
Number analyzed (Participants) | 48 | 2 | 12
scores on a scale | -2.3 (4.6) | 0.0 (0.0) | -0.3 (1.0)

31. Secondary Outcome: Certolizumab Pegol (CZP) Plasma Concentration During the Study
Description: CZP plasma concentration was measured in micrograms per milliliter (μg/mL). Blood sample measurements that were deemed to be below the level of quantification, were set to half the lower level of quantification (LLOQ) for analysis purposes. Summary statistics were only displayed if at least two-thirds of the values were above the LLOQ and if n was greater or equal to (>=) 4.
  The primary purpose of the study was to evaluate treatment options for axSpA patients after being in sustained remission. Hence, one of the objectives was to evaluate the PK of these patients. The CZP plasma concentration of the patients that did not reach sustained remission were therefore not analysed, and the Pharmacokinetic Set A as described in the protocol was removed from the SAP.
Time Frame: From Week 0 until the Safety Follow-up Visit (10 weeks after the last dose of study medication)
Population: The Pharmacokinetic Set B (PKSB) consisted of all study participants from the Safety Set Part B (SSB) who provided at least 1 PK sample during Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Placebo Double-Blind (PKSB): Participants in this arm received Placebo subcutaneous (sc) every 2 weeks from Week 48 onwards.
  Participants formed the Pharmacokinetic Set B (PKSB).
- Certolizumab Pegol 200 mg Q2W Double-Blind (PKSB): Participants in this arm received certolizumab pegol (CZP) 200 mg subcutaneous (sc) every 2 weeks (Q2W) from Week 48 onwards.
  Participants formed the PKSB.
- Certolizumab Pegol 200 mg Q4W Double-Blind (PKSB): Participants in this arm received certolizumab pegol (CZP) 200 mg subcutaneous (sc) every 4 weeks (Q4W) from Week 48 onwards. At visits where CZP was not received, subjects received one injection of Placebo to maintain the study blind.
  Participants formed the PKSB.
Arm/Group | Placebo Double-Blind (PKSB) | Certolizumab Pegol 200 mg Q2W Double-Blind (PKSB) | Certolizumab Pegol 200 mg Q4W Double-Blind (PKSB)
Number analyzed (Participants) | 101 | 102 | 105
μg/mL
  Part A Baseline: number analyzed (Participants) | 99 | 101 | 105
  Part A Baseline | NA (NA) — Participants had no prior CZP treatment and thus no CZP levels at Baseline. | NA (NA) — Participants had no prior CZP treatment and thus no CZP levels at Baseline. | NA (NA) — Participants had no prior CZP treatment and thus no CZP levels at Baseline.
  Week 4: number analyzed (Participants) | 101 | 100 | 104
  Week 4 | 48.71 (85.76) | 53.39 (30.93) | 48.92 (43.17)
  Week 12: number analyzed (Participants) | 100 | 101 | 105
  Week 12 | 30.91 (89.23) | 31.74 (50.79) | 30.69 (56.82)
  Week 24: number analyzed (Participants) | 100 | 101 | 104
  Week 24 | 26.31 (135.58) | 30.23 (46.57) | 28.96 (58.38)
  Week 48/Part B Baseline: number analyzed (Participants) | 98 | 100 | 104
  Week 48/Part B Baseline | 36.28 (74.18) | 36.59 (84.36) | 31.11 (138.29)
  Week 60: number analyzed (Participants) | 98 | 100 | 105
  Week 60 | NA (NA) — Values were below the level of detection. | 27.76 (49.47) | 6.95 (178.27)
  Week 72: number analyzed (Participants) | 76 | 95 | 99
  Week 72 | NA (NA) — Values were below the level of detection. | 26.36 (105.58) | 7.61 (176.39)
  Week 84: number analyzed (Participants) | 38 | 91 | 90
  Week 84 | NA (NA) — Values were below the level of detection. | 26.57 (44.90) | 8.00 (113.48)
  Week 96: number analyzed (Participants) | 27 | 86 | 85
  Week 96 | NA (NA) — Values were below the level of detection. | 24.76 (97.60) | 7.16 (131.76)
  Withdrawal Visit: number analyzed (Participants) | 4 | 3 | 5
  Withdrawal Visit | 0.81 (1802.40) | NA (NA) — Values were below the level of detection. | 0.30 (2621.06)
  Escape Week 0/Flare Baseline: number analyzed (Participants) | 72 | 6 | 14
  Escape Week 0/Flare Baseline | NA (NA) — Values were below the level of detection. | 30.77 (19.78) | 12.70 (98.45)
  Escape Week 2: number analyzed (Participants) | 71 | 6 | 15
  Escape Week 2 | 18.27 (488.45) | 33.50 (21.17) | 15.43 (124.10)
  Escape Week 4: number analyzed (Participants) | 71 | 6 | 15
  Escape Week 4 | 37.32 (151.18) | 32.94 (30.48) | 18.43 (79.93)
  Escape Week 12: number analyzed (Participants) | 69 | 6 | 15
  Escape Week 12 | 23.89 (232.36) | 23.76 (65.42) | 19.14 (136.22)
  Escape Week 24: number analyzed (Participants) | 54 | 3 | 8
  Escape Week 24 | 27.47 (45.31) | NA (NA) — Values were below the level of detection. | 19.23 (66.68)
  Escape Week 36: number analyzed (Participants) | 14 | 3 | 3
  Escape Week 36 | 24.88 (77.53) | NA (NA) — Values were below the level of detection. | NA (NA) — Values were below the level of detection.
  Last Visit (Week 96): number analyzed (Participants) | 66 | 6 | 14
  Last Visit (Week 96) | 24.64 (112.75) | 26.19 (54.74) | 18.59 (95.75)
  Withdrawal Escape Visit: number analyzed (Participants) | 4 | 1 | 0
  Withdrawal Escape Visit | 4.71 (133329.3) | NA (NA) — Values were below the level of detection. |
  Safety Follow-up: number analyzed (Participants) | 92 | 92 | 98
  Safety Follow-up | NA (NA) — Values were below the level of detection. | 0.52 (1158.85) | 0.14 (772.54)

32. Secondary Outcome: Percentage of Participants With Positive Anti-certolizumab Pegol-antibody Levels in Plasma During the Study
Description: Treatment emergent ADAb status positive was defined as either baseline ADAb negative subjects having at least one ADAb confirmed positive sample post baseline or baseline ADAb positive subjects with at least one post baseline sample with >= minimum significant ratio (MSR) increase from baseline on CZP treatment. Once determined positive, the highest titer during Part A and Part B (including Escape and Safety Follow up) was used to categorize the subject.
  The primary purpose of the study was to evaluate treatment options for axSpA patients after being in sustained remission. Hence, one of the objectives was to evaluate the immunogenicity of these patients. The ADAb titer of the patients that did not reach sustained remission were therefore not analysed, and the Pharmacokinetic Set A as described in the protocol was removed from the SAP.
Time Frame: From Week 0 until the Safety Follow-up Visit (10 weeks after the last dose of study medication)
Population: as for outcome 31
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Double-Blind (PKSB) | Certolizumab Pegol 200 mg Q2W Double-Blind (PKSB) | Certolizumab Pegol 200 mg Q4W Double-Blind (PKSB)
Number analyzed (Participants) | 101 | 102 | 105
percentage of participants | 100 | 96.1 | 100

33. Secondary Outcome: Percentage of Participants With at Least One Adverse Event (AE) During Part A of the Study
Description: An AE was any untoward medical occurrence in a patient or clinical investigation study participant administered a pharmaceutical product that did not necessarily have a causal relationship with this treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From Screening Period (Week -5 to Week -1) until Week 48
Population: The Safety Set (SS) consisted of all study participants in the Enrolled Set (ES) who received at least 1 dose of investigational medicinal product (IMP).
Measure: Number; unit: percentage of participants
Groups:
- Certolizumab Pegol Open-Label (SS) Wk 0-48: Participants in this arm received certolizumab pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 6 to Week 48 (Part A). Participants in sustained remission at Week 48 were eligible for randomization into Part B.
  Participants formed the Safety Set (SS).
Arm/Group | Certolizumab Pegol Open-Label (SS) Wk 0-48
Number analyzed (Participants) | 736
percentage of participants
  Screening Period (Week -5 to Week -1) | 7.3
  Open-Label Period (Week 0 to Week 48) | 67.9

34. Secondary Outcome: Percentage of Participants With at Least One Adverse Event (AE) During Part B of the Study
Description: An AE was any untoward medical occurrence in a patient or clinical investigation study participant administered a pharmaceutical product that did not necessarily have a causal relationship with this treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
  For subjects with flare in Part B and do escape to CZP full-dose therapy, only TEAEs with an onset date prior to the start date of escape CZP full-dose therapy were included.
Time Frame: From Week 0 until the Safety Follow-up Visit (10 weeks after the last dose of study medication)
Population: The Safety Set Part B (SSB) consisted of all study participants in the Randomized Set (RS) who received at least 1 dose of IMP in the Double-Blind Period of the study (Part B).
Measure: Number; unit: percentage of participants
Groups:
- Placebo Double-Blind (SSB) Wk 48-96: Participants in this arm received Placebo subcutaneous (sc) every 2 weeks from Week 48 onwards.
  Participants formed the Safety Set Part B (SSB).
- Certolizumab Pegol 200 mg Q2W Double-Blind (SSB) Wk 48-96: Participants in this arm received certolizumab pegol (CZP) 200 mg subcutaneous (sc) every 2 weeks (Q2W) from Week 48 onwards.
  Participants formed the SSB.
- Certolizumab Pegol 200 mg Q4W Double-Blind (SSB) Wk 48-96: Participants in this arm received certolizumab pegol (CZP) 200 mg subcutaneous (sc) every 4 weeks (Q4W) from Week 48 onwards. At visits where CZP was not received, subjects received one injection of Placebo to maintain the study blind.
  Participants formed the SSB.
Arm/Group | Placebo Double-Blind (SSB) Wk 48-96 | Certolizumab Pegol 200 mg Q2W Double-Blind (SSB) Wk 48-96 | Certolizumab Pegol 200 mg Q4W Double-Blind (SSB) Wk 48-96
Number analyzed (Participants) | 103 | 104 | 105
percentage of participants | 54.4 | 57.7 | 61.0

35. Secondary Outcome: Percentage of Participants With at Least One Adverse Event (AE) and Who Experienced a Flare During Part B of the Study
Description: An AE was any untoward medical occurrence in a patient or clinical investigation study participant administered a pharmaceutical product that did not necessarily have a causal relationship with this treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
  For subjects with flare in Part B and do escape to CZP full-dose therapy, only TEAEs with an onset date after or on the start date of escape CZP full-dose therapy were included.
Time Frame: From time of flare to Escape Week 12
Population: The Escape Therapy Set (ETS) consisted of all study participants from the Flared Set (FS) who received at least 1 dose of escape treatment.
Measure: Number; unit: percentage of participants
Groups:
- Placebo DB/CZP 200 mg Q2W Escape (ETS) Escape Wk 0->=12: Participants randomized to Placebo who met flare criteria received CZP 400 mg subcutaneous (sc) every 2 weeks (Q2W) for the first 3 visits after flare has been confirmed. After that, CZP 200 mg was given every 2 weeks in open-label fashion. The duration was from starting escape treatment after flare until Week 96 with a minimum of 12 weeks.
  Participants formed the Escape Therapy Set (ETS).
- CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (ETS) Escape Wk 0->=12: Participants randomized to CZP 200 mg Q2W who meet flare criteria received CZP 200 mg subcutaneous (sc) every 2 weeks (Q2W) for all visits after flare has been confirmed. At the first 3 visits after flare has been confirmed, participants received one injection of 200 mg CZP and one injection of Placebo to maintain the study blind. The duration was from starting escape treatment after flare until Week 96 with a minimum of 12 weeks.
  Participants formed the ETS.
- CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (ETS) Escape Wk 0->=12: Participants randomized to CZP 200 mg Q4W who meet flare criteria received CZP 200 mg subcutaneous (sc) every 2 weeks (Q2W) for all visits after flare has been confirmed. At the first 3 visits after flare has been confirmed, participants received one injection of 200 mg CZP and one injection of Placebo to maintain the study blind. The duration was from starting escape treatment after flare until Week 96 with a minimum of 12 weeks.
  Participants formed the ETS.
Arm/Group | Placebo DB/CZP 200 mg Q2W Escape (ETS) Escape Wk 0->=12 | CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (ETS) Escape Wk 0->=12 | CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (ETS) Escape Wk 0->=12
Number analyzed (Participants) | 72 | 6 | 15
percentage of participants | 51.4 | 83.3 | 46.7

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Week 0 (Baseline) until the Safety Follow-Up Period (10 weeks after the last dose of study medication).
Description: TEAEs counts are for each study period: Open-Label (Wk0-48), Double-Blind (Wk48-96) and Escape (Wk0-12). During Escape (last 3 columns) all participants received CZP 200 mg Q2W at time of TEAEs, although they were coming from 3 arms of the double-blind phase. Participants randomized or who entered escape but received no treatment are not included.
Arm/Group | Certolizumab Pegol Open-Label (SS) Wk 0-48 | Placebo Double-Blind (SSB) Wk 48-96 | Certolizumab Pegol 200 mg Q2W Double-Blind (SSB) Wk 48-96 | Certolizumab Pegol 200 mg Q4W Double-Blind (SSB) Wk 48-96 | Placebo DB/CZP 200 mg Q2W Escape (ETS) Escape Wk 0->=12 | CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (ETS) Escape Wk 0->=12 | CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (ETS) Escape Wk 0->=12
All-Cause Mortality (participants affected / at risk) | 0/736 | 0/103 | 0/104 | 0/105 | 0/72 | 0/6 | 0/15
Serious Adverse Events (participants affected / at risk) | 44/736 | 0/103 | 5/104 | 0/105 | 0/72 | 1/6 | 0/15
Other Adverse Events (participants affected / at risk) | 188/736 | 25/103 | 31/104 | 26/105 | 20/72 | 5/6 | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol Open-Label (SS) Wk 0-48 (N=736) | Placebo Double-Blind (SSB) Wk 48-96 (N=103) | Certolizumab Pegol 200 mg Q2W Double-Blind (SSB) Wk 48-96 (N=104) | Certolizumab Pegol 200 mg Q4W Double-Blind (SSB) Wk 48-96 (N=105) | Placebo DB/CZP 200 mg Q2W Escape (ETS) Escape Wk 0->=12 (N=72) | CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (ETS) Escape Wk 0->=12 (N=6) | CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (ETS) Escape Wk 0->=12 (N=15)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tuberculous pleurisy (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
False positive tuberculosis test (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axial spondyloarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Latent tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol Open-Label (SS) Wk 0-48 (N=736) | Placebo Double-Blind (SSB) Wk 48-96 (N=103) | Certolizumab Pegol 200 mg Q2W Double-Blind (SSB) Wk 48-96 (N=104) | Certolizumab Pegol 200 mg Q4W Double-Blind (SSB) Wk 48-96 (N=105) | Placebo DB/CZP 200 mg Q2W Escape (ETS) Escape Wk 0->=12 (N=72) | CZP 200 mg Q2W DB/CZP 200 mg Q2W Escape (ETS) Escape Wk 0->=12 (N=6) | CZP 200 mg Q4W DB/CZP 200 mg Q2W Escape (ETS) Escape Wk 0->=12 (N=15)
Nasopharyngitis (Infections and infestations) | 117 (156) | 8 (8) | 12 (17) | 13 (18) | 8 (9) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 63 (88) | 10 (12) | 12 (14) | 11 (12) | 5 (7) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 22 (24) | 3 (3) | 2 (2) | 6 (6) | 2 (2) | 0 (0) | 1 (1)
Axial spondyloarthritis (Musculoskeletal and connective tissue disorders) | 8 (8) | 8 (8) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 8 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oral herpes (Infections and infestations) | 13 (21) | 2 (3) | 1 (3) | 2 (2) | 1 (1) | 1 (3) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 9 (9) | 1 (1) | 3 (3) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 24 (25) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 6 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Latent tuberculosis (Infections and infestations) | 5 (5) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 12 (12) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Antinuclear antibody increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervicogenic vertigo (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT02505542/SAP_000.pdf
  • Study Protocol (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT02505542/Prot_001.pdf